CLINICAL TRIAL: NCT04447144
Title: Nutritional Habits, Does it Affect Coronavirus Disease 2019 (COVID-19) Infection Outcome? An Egyptian Experience
Brief Title: Nutritional Habits, and Coronavirus Disease 2019 (COVID-19) Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Hegazy, Professor of Internal Medicine Hepatology & gastroenterology Unit Faculty of medicine, Cairo University, Cairo University, Cairo University
Other Study IDs: 1003
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Covid19; Chronic Inflammation; Non-Communicable Chronic Diseases
Keywords: Covid19; noncommunicable diseases; chronic inflammation; Mediterranean diet
MeSH Terms: conditions — COVID-19; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 mild severity: Definition of mild cases according to MOH:
  1. Age < 60
  2. Temperature <38.5
  3. arterial oxygen saturation (SaO2) >92%
  4. Heart Rate <110
  5. Respiratory Rate <25 /min.
  6. Neutrophil / lymphocyte ratio on complete blood count (CBC) < 3.1
  7. No co-morbidities that necessitates hospital admission: Pregnancy, severe uncontrolled Diabetes, Chronic lung disease, Chronic kidney disease, Chronic liver disease, Serious heart diseases (arrythmia, Ischemic heart disease, uncontrolled hypertension), immunocompromised: prolonged use of corticosteroids and other immunosuppressive drugs/ organ transplantation/ HIV/ Immunodeficiency, Obesity (BMI > 40)
- COVID-19 moderate severity: Any patient not fulfilling the above mild criteria is considered having moderate disease as well as any positive pulmonary imaging findings

SUMMARY:
As of May 30th more than 23,000 cases of COVID -19 cases were confirmed in Egypt with total deaths of 913. Post viral entry, intense immune response against the virus with infiltration of monocytes and macrophages into alveolar cells with decreasing number of lymphocytes in peripheral blood along with reduced lymphocytes in lymphoid organs, hypercoagulability, thrombosis and multiple organ damage, The gut microbiota and immune homeostasis seem to have a back and forth relationship.

Also, gut microbiota derived signals are known to tune the immune cells for pro and anti-inflammatory responses thereby affecting the susceptibility to various diseases. Healthy gut microbiome essentially could be pivotal in maintaining an optimal immune system to prevent an array of excessive immune reactions that eventually become detrimental to lungs and vital organ systems.

Numerous studies have shown that the patient's nutritional status have a significant effect on an individual's immunity and over all health status and it has been suggested that nutritional deficiencies may predispose to severe forms of COVID-19 infections.

Co-existing non-communicable chronic diseases (NCDs) in COVID-19 patients have been found to delay patients recovery and worsen their prognosis, the reason may be due to aggravated inflammatory pathology found in NCDs exacerbating COVID-19 infection.

The aim of the study is to evaluate the role dietary habits among COVID-19 Egyptian patients and whether type of diet (Mediterranean or Western) will affect disease outcomes

DETAILED DESCRIPTION:
As of May 30th more than 23,000 cases of COVID -19 cases were confirmed in Egypt with total deaths of 913. There are over six million confirmed cases of COVID-19 and almost 370,000 deaths globally. COVID-19 originated from Wuhan city, China in early 2020, from their extending to the rest of the world. The virus belong to a large class of viruses known as β-coronaviruses with a large number of potential natural primary, intermediate and final hosts. Severe acute respiratory syndrome corona virus 2 (SARS-CoV-2) is an enveloped RNA virus that typically spread by droplets causing pulmonary and extra-pulmonary complications.

COVID-19 can result in cytokine storm, which in severe cases can lead to acute respiratory distress syndrome (ARDS), sepsis and multiple organ dysfunction that can progress to death. Post SARS-CoV-2 entry, intense immune response against the virus with infiltration of monocytes and macrophages into alveolar cells with decreasing number of lymphocytes in peripheral blood along with reduced lymphocytes in lymphoid organs, hypercoagulability, thrombosis and multiple organ damage. This along with the fact that some patients of this disease have diarrhea points out towards a distinct possibility of involvement of gut-lung axis and may be the gut microbiota.

The gut microbiota and immune homeostasis seem to have a back and forth relationship. Also, gut microbiota derived signals are known to tune the immune cells for pro and anti-inflammatory responses thereby affecting the susceptibility to various diseases.

Many elderly and immune-compromised patients progress to serious adverse clinical outcomes, it is therefore tempting to speculate that in COVID-19, there is a possible cross-talk taking place between the lung and the gut microbiota which might influence the outcome of the clinical manifestation.

Healthy gut microbiome essentially could be pivotal in maintaining an optimal immune system to prevent an array of excessive immune reactions that eventually become detrimental to lungs and vital organ systems.

Several studies have shown that increased D-dimer levels are associated with severe forms of COVID-19 infection, this might be explained by diffuse alveolar damage, pneumocytes desquamation, pulmonary edema, interstitial mononuclear cells and lymphocytes infiltration causing intense inflammatory burden induced in severe COVID-19 infections.

Numerous studies have shown that the patient's nutritional status have a significant effect on an individual's immunity and over all health status and it has been suggested that nutritional deficiencies may predispose to severe forms of COVID-19 infections. Adequate Fruits and vegetables consumption have been studied for their potential protective effects against respiratory diseases and anti-inflammatory effects, furthermore, fruits and vegetables are also rich sources of fibers that have favorable effects on gut microbiome. One of very familiar water-soluble vitamins; Vitamin C (ascorbic acid) , that can be found in citrus fruits, barriers, leafy greens, tomatoes, and various other fruits and vegetables. Indeed, 1-2 g supplementation of vitamin C was found to shorten the duration of common cold by 18%, according to the United states National Institute of health (NIH) the recommended daily allowances (RDA) of vitamin C for healthy adults is 75-90 mg/d.

The Sunshine vitamin (Vitamin D) which is found in mushrooms, eggs, salmon and milk was found in a meta-analysis of 25 randomized controlled trails conducted over more than 11,000 participants, an overall protective effect of vitamin D supplementation in acute respiratory infections and, also, COVID-19, studies also suggested to possible role of Vitamin D as an antiviral immunomodulator through anti-inflammatory properties, for this reason, Vitamin D have been suggested to have a beneficial effects against SARS-CoV-2 infection (16), another study done in Switzerland on SARS-CoV-2 positive patients found to have significant lower levels (mean value 11.1 ng/mL) of 25-hydroxyvitamin D. The recommended RDA of vitamin D according to NIH 15-20 ug/d (600-800 IU with tolerable upper limit of 4000 IU). Another vitamin with anti-inflammatory benefits, fat soluble vitamin E (œ-tocopherol) found in seeds, green leafy vegetables, nuts, and fortified cereals. Vitamin E has been labeled as immunoenhancing vitamin by with anti-inflammatory properties by regulating the production of Reactive Oxygen Species (ROS) and Reactive Nitrogen Species (RNS) and modulating signal transduction, thus protecting The polyunsaturated fatty acids (PUFAs) in the cell membranes, for this reason, it has been suggested that the combination of Vitamins C, D & E may be useful in COVID-19 patients. The RDA of Vitamin E for healthy adults according to the NIH is 15 mg/d (tolerable upper level 1000 mg/d).

Regarding minerals, Zinc has been found to have a critical role in maintaining immune cells integrity and important cofactor for numerous enzyme, zinc deficiency can cause impaired cell-mediated immunity predisposing to various infections, especially respiratory infections, available food sources of zinc including; meats, legumes and diary products, the RDA of zinc according to NIH is 8-11 mg/d (with 40 mg/day tolerable upper intake level).

Another essential trace element is Copper that can be found in nuts and offal and, in lesser concentrations in cereals and fruits, copper has a pivotal role in maintaining DNA integrity by its antioxidant effects, studies have shown that adequate copper supplementation can reduce lung inflammation in mice, according to NIH, the RDA of copper is 900 ug/d (tolerable upper limit of 10 mg/d).

Regular intake of prebiotic foods such as oligosaccharides, fermentable fibers, and resistant starches can beneficially affect the gut microbiota, prebiotic fibers are considered selective substrates for specific beneficial colonic bacteria as they are neither hydrolyzed nor absorbed in the proximal gut. Dietary fibers have been suggested as immunity modulators as they lower incidence of bacterial translocation by maintaining integrity of the gut barrier, available sources include; oat, barley, seeds, nuts, peas and some fruits, the recommended daily intake is 25-38 g/day. Probiotic foods (from dairy products as yogurt& sour cream) and supplements have the ability to modify the gut microbiota and potentially modulate gut inflammatory response.

D-dimer is a fibrin degradation product (FDP) that reflects bath thrombin production and activation, elevated levels have been linked to increased risk of coronary artery disease, cerebrovascular strokes and total mortality, so far the link between dietary habits and D-dimer levels has been poorly explored. Studies have reported, that adherence to a Mediterranean diet was found to be associated with decreased levels of D-dimer, with possible antithrombotic effects due to high content of fibers, antioxidants, mono and polyunsaturated fatty acids.

Co-existing non-communicable chronic diseases (NCDs) in COVID-19 patients have been found to delay patients recovery and worsen their prognosis, the reason may be due to aggravated inflammatory pathology found in NCDs exacerbating COVID-19 infection. Such patients with underlying cardiovascular, respiratory disease were found to have worse prognosis, diabetes, hypertension and hypercholesterolemia are considered major risk factors for thrombotic complications, which in COVID-19 patients may account for higher risk of serious disease outcome and is associated with two-folds increase in mortality.

Fish and fish oils are considered very beneficial to individual health especially in patients with NCDs including cardiovascular diseases. Omega-3-polyunsaturated fatty acids (PUFA) are integral component of the cell membrane thus having anti-inflammatory effects, however, substantial human trials in this area are lacking.

For this reason, an effective approach to reduce person's risk of developing NCDs is to halt underlying inflammation via modifiable risk factors including; diet, exercise and healthy lifestyle choices. To date, there is no single food or natural remedy that has been used for preventing COVID-19 infections. Healthy diets containing adequate amounts of necessary macro and micronutrients, prebiotics and probiotics that can maintain and restore immune system, therefore increasing protection against chronic inflammation-related NCDs. Foods with anti-inflammatory and immunomodulatory compounds including essential vitamins (C, D & E) and minerals (Zinc, Copper, Calcium & Selenium) are considered protective foods, these micronutrients can act in harmony to prevent thrombotic and reactive oxygen species (ROS) complications by their anti-inflammatory properties. They are present in fair amounts in Mediterranean Diet, which is characterized by increased dietary consumption of legumes, olive oil, whole grains, nuts, and monounsaturated fats, minimally processed fruits, vegetables, associated with low to moderate consumption of fermented dairy products, fish, poultry. Antithrombotic advantages of Mediterranean diet have been explained by reduced levels of factor VII, tissue factor, platelets and leucocytes counts in individuals consuming Mediterranean diet. On the other hand, The "Western" dietary pattern, which is characterized by high consumption of saturated fats, refined carbohydrates, red meat, deserts and sweets, that may be associated with hyperglycemia, hyperlipidemia and chronic inflammatory state.

The aim of the study is to evaluate the role dietary habits among COVID-19 Egyptian patients and whether type of diet (Mediterranean or Western) will affect disease outcomes.

The current study also trying to determine if balanced diet maintaining healthy gut microbiota can have a role in avoiding disease progression and deterioration in COVID-19 cases.

Dietary pattern questionnaire for COVID 19 patient Name:- Age :- The work:- height :- Weight :- BMI :-

* Did you lose weight during the previous 3 months?
* Do you smoke?
* What is your usual breakfast before the injury and when to take it ?
* What is your usual lunch before the injury and when to take it ?
* What is your usual dinner before the injury and when to take it ?
* Did you eat between meals and what you eat?
* How many cups of water you drink daily?
* Do you eat salads or fresh vegetables daily (type and amount)?
* Do you eat fruit daily (type and amount )?
* Do you drink milk daily ?
* Do you eat yogurt daily?
* Do you drink fermented milk daily?
* Do you eat cheese daily(type and amount)?
* Do you eat fish weekly ( type and amount)?
* Do you eat pickles daily(amount) ?
* Are you exposed to the sun daily ( duration and time)?
* Number of spoons of sugar taken per day ( and sweets)?
* Types of drinks daily and their times ?
* Frequency of eating out ( weekly)?
* Do you eat any of these food daily ( cocoa , cashew , cheddar, chicken , meat, Milk , almond , salmon , yogurt)?
* Number of times eating eggs per week ?
* The type and amount of fats used in cooking :-
* Number of hours of sleep per day :-
* Antibiotic intake rate:-
* Have you take any supplements and vitamins for the past months?

The analysis of the above food habits questionnaire Will be fitted to a scoring system from 0 to 32 points covering the following

1. Probiotic in food
2. Prebiotic in food
3. Vitamins and minerals in food
4. Mediterranean type of food
5. Antibiotics intake that affect gut microbiota
6. Tea frequency and amount intake with respecting it's role on microbiota
7. Exercise daily and it's effect on immune system and lung capacity

All patients will be followed up for 14 days For disease recovery or progression to severe category.

Statistical analysis will be done after tabulation of the results to correlate with microbiome as well as the clinical status of patients.

Aim and Expected outcomes: The novelty of this study is that the investigators will get information about the role and type of diet on COVID-19 outcome and clarifying the role certain macro and micronutrients in inducing chronic inflammation, protecting from thrombosis The investigators also hope through this research to modify dietary habits in the Egyptian society encouraging healthy nutrition with the pre and probiotics food role to retain normal healthy life.

ELIGIBILITY:
Inclusion Criteria:

- Patients (18 -80 years) with mild to moderate COVID-19 cases consented to home or hospital isolation to follow them.

Exclusion Criteria:

Severe cases not fulfilling the definition of mild and moderate cases.

Definition of mild cases according to The Egyptian Ministry Of Health: (MOH)

1. Age < 60
2. Temperature <38.5
3. SaO2 >92%
4. Heart Rate <110
5. Respiratory Rate <25 /min.
6. Neutrophil / lymphocyte ratio on CBC < 3.1
7. No co-morbidities that necessitates hospital admission: Pregnancy, severe uncontrolled Diabetes, Chronic lung disease, Chronic kidney disease, Chronic liver disease, Serious heart diseases (arrythmia, Ischemic heart disease, uncontrolled hypertension), immunocompromised: prolonged use of corticosteroids and other immunosuppressive drugs/ organ transplantation/ HIV/ Immunodeficiency, Obesity (BMI > 40) Any patient not fulfilling the above mild criteria is considered having moderate disease as well as any positive pulmonary imaging findings

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a prospective cross-sectional single center National study, will include 200 Egyptian patients. The patients preliminary suggested to have COVID-19 of mild to moderate severity that is confirmed by laboratory and imaging studies.
  Blood samples will be obtained for:
  * CBC including lymphocyte count and absolute neutrophil count
  * ALT, AST, bilirubin total and direct
  * Serum creatinine, urea
  * C- reactive protein
  * LDH
  * D-dimer
  * Serum ferritin 4. ECG, CXR & CT chest will be done and followed with Labs. 5. A questionnaire for the diet will be filled by the patient and will be analyzed.
    6. All patients will receive Hydroxychloroquine, Vitamin C, Zink tablets, acetylcysteine and lacorferrin according to The Egyptian Ministry of Health treatment protocol for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Western versus Mediterranean diet in COVID-19 outcome | 2 months
  To assess the relation between type of diet in mild to moderate COVID 19, to the fate of their course; either improvement or progression
Gut- Lung axis in COVID-19 | 2 months
  To asses any possible links between gut microbiome and the lung affecting clinical presentation of mild to moderate COVID cases; as diarrhea, loss of taste or smell
Protective role of minerals and vitamins in COVID-19 patients | 2 months
  Possible protective effects of minerals and vitamins against COVID-19 respiratory illness
non-communicable diseases and COVID-19 | 2 months
  Trying to explain the link between non-communicable disease severity and COVID-19 prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Abdul Ghani, MD, Study Director — Lecture of Internal Medicine Hepatology & gastroenterology Unit
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Egypt

REFERENCES:
- [Background] John Hopkins University. John Hopkins University & Medicine: Coronavirus Resource Center. Available online: https://coronavirus.jhu.edu/map.html
- [Background] Wang L, Wang Y, Ye D, Liu Q. Erratum to ;;A review of the 2019 Novel Coronavirus (COVID-19) based on current evidence'' [International Journal of Antimicrobial Agents 55/6 (2020) 105948]. Int J Antimicrob Agents. 2020 Sep;56(3):106137. doi: 10.1016/j.ijantimicag.2020.106137. Epub 2020 Aug 18. No abstract available. PMID 32826129
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Zhang W, Zhao Y, Zhang F, Wang Q, Li T, Liu Z, Wang J, Qin Y, Zhang X, Yan X, Zeng X, Zhang S. The use of anti-inflammatory drugs in the treatment of people with severe coronavirus disease 2019 (COVID-19): The Perspectives of clinical immunologists from China. Clin Immunol. 2020 May;214:108393. doi: 10.1016/j.clim.2020.108393. Epub 2020 Mar 25. PMID 32222466
- [Background] Chin VK, Yong VC, Chong PP, Amin Nordin S, Basir R, Abdullah M. Mycobiome in the Gut: A Multiperspective Review. Mediators Inflamm. 2020 Apr 4;2020:9560684. doi: 10.1155/2020/9560684. eCollection 2020. PMID 32322167
- [Background] Negi S, Pahari S, Bashir H, Agrewala JN. Gut Microbiota Regulates Mincle Mediated Activation of Lung Dendritic Cells to Protect Against Mycobacterium tuberculosis. Front Immunol. 2019 May 28;10:1142. doi: 10.3389/fimmu.2019.01142. eCollection 2019. PMID 31231363
- [Background] Nagpal R, Mainali R, Ahmadi S, Wang S, Singh R, Kavanagh K, Kitzman DW, Kushugulova A, Marotta F, Yadav H. Gut microbiome and aging: Physiological and mechanistic insights. Nutr Healthy Aging. 2018 Jun 15;4(4):267-285. doi: 10.3233/NHA-170030. PMID 29951588
- [Background] Round JL, Mazmanian SK. Inducible Foxp3+ regulatory T-cell development by a commensal bacterium of the intestinal microbiota. Proc Natl Acad Sci U S A. 2010 Jul 6;107(27):12204-9. doi: 10.1073/pnas.0909122107. Epub 2010 Jun 21. PMID 20566854
- [Background] Yao Y, Cao J, Wang Q, Shi Q, Liu K, Luo Z, Chen X, Chen S, Yu K, Huang Z, Hu B. D-dimer as a biomarker for disease severity and mortality in COVID-19 patients: a case control study. J Intensive Care. 2020 Jul 10;8:49. doi: 10.1186/s40560-020-00466-z. eCollection 2020. PMID 32665858
- [Background] Zhang L, Liu Y. Potential interventions for novel coronavirus in China: A systematic review. J Med Virol. 2020 May;92(5):479-490. doi: 10.1002/jmv.25707. Epub 2020 Mar 3. PMID 32052466
- [Background] Hemila H, Chalker E. Vitamin C for preventing and treating the common cold. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD000980. doi: 10.1002/14651858.CD000980.pub4. PMID 23440782
- [Background] Krinsky,N.I.; Beecher,G. ; Burk,R.; Chan,A.; Erdman,j.J.; Jacob,R.; Jialal,I.; Kolonel,L.; Marshall,J.;Taylor Mayne, P.R. Dietary Reference Intakes for Vitamin C, Vitamin E, Selenium, and Carotenoids; A Report of the Panel on Dietary Antioxidants and Related Compounds, Subcommittees on Upper Reference Levels of Nutrients and Interpretation and Uses of Dietary Reference Intakes, and the Standing Committee on the Scientific Evaluation of Dietary Reference Intakes, Institute of Medicine; The National Academies Press: Washington, DC, USA, 2000.
- [Background] Martineau AR, Jolliffe DA, Hooper RL, Greenberg L, Aloia JF, Bergman P, Dubnov-Raz G, Esposito S, Ganmaa D, Ginde AA, Goodall EC, Grant CC, Griffiths CJ, Janssens W, Laaksi I, Manaseki-Holland S, Mauger D, Murdoch DR, Neale R, Rees JR, Simpson S Jr, Stelmach I, Kumar GT, Urashima M, Camargo CA Jr. Vitamin D supplementation to prevent acute respiratory tract infections: systematic review and meta-analysis of individual participant data. BMJ. 2017 Feb 15;356:i6583. doi: 10.1136/bmj.i6583. PMID 28202713
- [Background] Grant WB, Lahore H, McDonnell SL, Baggerly CA, French CB, Aliano JL, Bhattoa HP. Evidence that Vitamin D Supplementation Could Reduce Risk of Influenza and COVID-19 Infections and Deaths. Nutrients. 2020 Apr 2;12(4):988. doi: 10.3390/nu12040988. PMID 32252338
- [Background] Teymoori-Rad M, Shokri F, Salimi V, Marashi SM. The interplay between vitamin D and viral infections. Rev Med Virol. 2019 Mar;29(2):e2032. doi: 10.1002/rmv.2032. Epub 2019 Jan 6. PMID 30614127
- [Background] Jakovac H. COVID-19 and vitamin D-Is there a link and an opportunity for intervention? Am J Physiol Endocrinol Metab. 2020 May 1;318(5):E589. doi: 10.1152/ajpendo.00138.2020. No abstract available. PMID 32297519
- [Background] D'Avolio A, Avataneo V, Manca A, Cusato J, De Nicolo A, Lucchini R, Keller F, Cantu M. 25-Hydroxyvitamin D Concentrations Are Lower in Patients with Positive PCR for SARS-CoV-2. Nutrients. 2020 May 9;12(5):1359. doi: 10.3390/nu12051359. PMID 32397511
- [Background] Institute of Medicine (US) Committee to Review Dietary Reference Intakes for Vitamin D and Calcium; Ross AC, Taylor CL, Yaktine AL, Del Valle HB, editors. Dietary Reference Intakes for Calcium and Vitamin D. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK56070/ PMID 21796828
- [Background] 19. Wu,D.; Meydani, S.N. Vitamin E ,immunity, and infection. In Nutrition, Immunity, and Infection; CRC Press: Boca Raton, FL, USA, 2017; pp. 197-212.
- [Background] Coquette A, Vray B, Vanderpas J. Role of vitamin E in the protection of the resident macrophage membrane against oxidative damage. Arch Int Physiol Biochim. 1986 Dec;94(5):S29-34. PMID 2440399
- [Background] Wang JZ, Zhang RY, Bai J. An anti-oxidative therapy for ameliorating cardiac injuries of critically ill COVID-19-infected patients. Int J Cardiol. 2020 Aug 1;312:137-138. doi: 10.1016/j.ijcard.2020.04.009. Epub 2020 Apr 6. No abstract available. PMID 32321655
- [Background] Prasad AS. Zinc in human health: effect of zinc on immune cells. Mol Med. 2008 May-Jun;14(5-6):353-7. doi: 10.2119/2008-00033.Prasad. PMID 18385818
- [Background] Hess SY, Lonnerdal B, Hotz C, Rivera JA, Brown KH. Recent advances in knowledge of zinc nutrition and human health. Food Nutr Bull. 2009 Mar;30(1 Suppl):S5-11. doi: 10.1177/15648265090301S102. PMID 19472599
- [Background] Lordan R, Tsoupras A, Mitra B, Zabetakis I. Dairy Fats and Cardiovascular Disease: Do We Really Need to be Concerned? Foods. 2018 Mar 1;7(3):29. doi: 10.3390/foods7030029. PMID 29494487
- [Background] Bost M, Houdart S, Oberli M, Kalonji E, Huneau JF, Margaritis I. Dietary copper and human health: Current evidence and unresolved issues. J Trace Elem Med Biol. 2016 May;35:107-15. doi: 10.1016/j.jtemb.2016.02.006. Epub 2016 Mar 5. PMID 27049134
- [Background] Uriu-Adams JY, Keen CL. Copper, oxidative stress, and human health. Mol Aspects Med. 2005 Aug-Oct;26(4-5):268-98. doi: 10.1016/j.mam.2005.07.015. PMID 16112185
- [Background] Liu L, Geng X, McDermott J, Shen J, Corbin C, Xuan S, Kim J, Zuo L, Liu Z. Copper Deficiency in the Lungs of TNF-alpha Transgenic Mice. Front Physiol. 2016 Jun 14;7:234. doi: 10.3389/fphys.2016.00234. eCollection 2016. PMID 27378943
- [Background] Arrieta,M.C.; Meddings,J.; Field,C.J. The immunomodulatory effects of dietary fiber and prebiotics in the gastrointestinal tract. In Non digestible Carbohydrates and Digestive Health; Paeschke, T.M., Aimutis, W.R., Eds.; Blackwell Publishing Ltd. and Institute of Food Technologists: Ames, IA, USA, 2011; pp. 37-77.
- [Background] Schley PD, Field CJ. The immune-enhancing effects of dietary fibres and prebiotics. Br J Nutr. 2002 May;87 Suppl 2:S221-30. doi: 10.1079/BJNBJN/2002541. PMID 12088522
- [Background] King DE, Mainous AG 3rd, Lambourne CA. Trends in dietary fiber intake in the United States, 1999-2008. J Acad Nutr Diet. 2012 May;112(5):642-8. doi: 10.1016/j.jand.2012.01.019. Epub 2012 Apr 25. PMID 22709768
- [Background] Hasan N, Yang H. Factors affecting the composition of the gut microbiota, and its modulation. PeerJ. 2019 Aug 16;7:e7502. doi: 10.7717/peerj.7502. eCollection 2019. PMID 31440436
- [Background] Di Castelnuovo A, Bonaccio M, De Curtis A, Costanzo S, Persichillo M, de Gaetano G, Donati MB, Iacoviello L; MOLI-SANI investigators. Higher adherence to the Mediterranean diet is associated with lower levels of D-dimer: findings from the MOLI-SANI study. Haematologica. 2017 Feb;102(2):e61-e64. doi: 10.3324/haematol.2016.156331. Epub 2016 Oct 20. No abstract available. PMID 27846616
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Wadman M, Couzin-Frankel J, Kaiser J, Matacic C. A rampage through the body. Science. 2020 Apr 24;368(6489):356-360. doi: 10.1126/science.368.6489.356. No abstract available. PMID 32327580
- [Background] Kumar A, Arora A, Sharma P, Anikhindi SA, Bansal N, Singla V, Khare S, Srivastava A. Is diabetes mellitus associated with mortality and severity of COVID-19? A meta-analysis. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):535-545. doi: 10.1016/j.dsx.2020.04.044. Epub 2020 May 6. PMID 32408118
- [Background] Moro K, Nagahashi M, Ramanathan R, Takabe K, Wakai T. Resolvins and omega three polyunsaturated fatty acids: Clinical implications in inflammatory diseases and cancer. World J Clin Cases. 2016 Jul 16;4(7):155-64. doi: 10.12998/wjcc.v4.i7.155. PMID 27458590
- [Background] Lordan R, Tsoupras A, Zabetakis I. Phospholipids of Animal and Marine Origin: Structure, Function, and Anti-Inflammatory Properties. Molecules. 2017 Nov 14;22(11):1964. doi: 10.3390/molecules22111964. PMID 29135918
- [Background] Yu E, Malik VS, Hu FB. Cardiovascular Disease Prevention by Diet Modification: JACC Health Promotion Series. J Am Coll Cardiol. 2018 Aug 21;72(8):914-926. doi: 10.1016/j.jacc.2018.02.085. PMID 30115231
- [Background] Phillips CM, Chen LW, Heude B, Bernard JY, Harvey NC, Duijts L, Mensink-Bout SM, Polanska K, Mancano G, Suderman M, Shivappa N, Hebert JR. Dietary Inflammatory Index and Non-Communicable Disease Risk: A Narrative Review. Nutrients. 2019 Aug 12;11(8):1873. doi: 10.3390/nu11081873. PMID 31408965
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Martinez-Gonzalez MA, Bes-Rastrollo M. Dietary patterns, Mediterranean diet, and cardiovascular disease. Curr Opin Lipidol. 2014 Feb;25(1):20-6. doi: 10.1097/MOL.0000000000000044. PMID 24370845
- [Background] Bonaccio M, Di Castelnuovo A, De Curtis A, Costanzo S, Persichillo M, Donati MB, Cerletti C, Iacoviello L, de Gaetano G; Moli-sani Project Investigators. Adherence to the Mediterranean diet is associated with lower platelet and leukocyte counts: results from the Moli-sani study. Blood. 2014 May 8;123(19):3037-44. doi: 10.1182/blood-2013-12-541672. Epub 2014 Mar 31. PMID 24687087
- [Background] Van Hylckama Vlieg A, Callas PW, Cushman M, Bertina RM, Rosendaal FR. Inter-relation of coagulation factors and d-dimer levels in healthy individuals. J Thromb Haemost. 2003 Mar;1(3):516-22. doi: 10.1046/j.1538-7836.2003.00080.x. PMID 12871460
- [Background] Varraso R, Fung TT, Barr RG, Hu FB, Willett W, Camargo CA Jr. Prospective study of dietary patterns and chronic obstructive pulmonary disease among US women. Am J Clin Nutr. 2007 Aug;86(2):488-95. doi: 10.1093/ajcn/86.2.488. PMID 17684223
- [Background] Sergi D, Boulestin H, Campbell FM, Williams LM. The Role of Dietary Advanced Glycation End Products in Metabolic Dysfunction. Mol Nutr Food Res. 2021 Jan;65(1):e1900934. doi: 10.1002/mnfr.201900934. Epub 2020 Apr 20. PMID 32246887
- [Derived] Hegazy MA, Fouad MM, Abd Elshafy SA, Abdelfatah D, Lithy RM, Abdelghani A, Ashoush OA. Beneficial role of healthy eating Index-2015 score & physical activity on COVID-19 outcomes. BMC Nutr. 2023 Oct 2;9(1):113. doi: 10.1186/s40795-023-00727-8. PMID 37784193